CLINICAL TRIAL: NCT01280201
Title: A Phase II, Open Label, Uncontrolled and Multicenter Trial of Pazopanib Given as a Single Agent in Patients With Progressive Advanced/Metastatic Neuroendocrine Tumors (NET): a Search for Activity, Safety, and Predictive Biomarkers
Brief Title: Pazopanib as Single Agent in Advanced NETs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE-1002; 2010-020749-28 (EudraCT Number)
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Results first posted 2019-03-04 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Advanced/Metastatic Neuroendocrine Tumors
Keywords: Neuroendocrine Tumors; Pazopanib; GETNE; Biomarkers
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pazopanib (Experimental)
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib — Single arm of pazopanib 800 mg (2x400mg) given once daily as a single agent.

SUMMARY:
The incidence of new diagnosed patients with NET of the digestive tract including carcinoid and pancreatic islet cells tumors ranges from 2 to 10 per 100,000 in the western Countries (Kulke M, Mayer R. N Engl J Med 340:858-868, 1999). Despite of the low incidence, the prevalence of these tumors is high because of their relatively long survival estimated in 35% at 5 years for those patients with well or moderate differentiated tumors (Yao JC, et al. J Clin Oncol. 2008;26:3063-3072). In fact, digestive NETs are the second most prevalent tumors derived from the digestive tract after colorectal carcinoma.

NETs are characterized by abundant vasculature, moreover VEGFR and VEGFR are overexpressed in 60-84% of the carcinoids and pancreatic islet cells NETs (Zhang et al. Cancer 2007;109:1478-1486). Other pro-angiogenic factors like the platelet derived growth factor (PDGFR) have been also involved in NET progression and development (Chaudhry A, et al.Cancer Res 1992;52:1006-12).

Pazopanib is an oral tyrosine kinase inhibitor of the VEGFR, PDGFR and KIT with a dual activity both as an antiangiogenic and also and anti-tumoral agent (Kumar et al. Mol Cancer Ther2007;6:2012-2021, Hurwitz et al. Clin Cancer Res 2009;15:4220-4227). Pazopanib seems to have a better toxicity profile versus the other antiangiogenic tyrosine kinase inhibitors and has already shown activity in several tumor types like renal cell carcinoma (Sternberg et al. J Clin Oncol 2009;27:abst. 5021), soft tissue sarcomas (Sleijfer et al. J Clin Oncol 2009;27:3126-32), hepatocellular carcinoma (Yau et al. J Clin Oncol 2009;27:abst. 3561), colorectal cancer (Brady et al. J Clin Oncol 2009;27:abst.4133), and thyroid cancers (Bible et al. J Clin Oncol 2009;27:abst. 3521).

The Spanish Group for Research in Neuroendocrine Tumors (GETNE) group is an active Member inside of the GENET group and has a large tradition in clinical trials in NETs. The investigators hypothesize that pazopanib may have at least as good activity and better safety profile than other VEGFR inhibitors in progressive advanced or metastatic NET tumors derived from the digestive tract.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must provide signed informed consent form prior to performance of study-specific procedures or assessments, and must be willing to comply with treatment and follow-up.

   Procedures conducted as part of the subject's clinical routine (e.g., blood count, imaging study) and obtained prior to signing the consent form might be used for screening or baseline purposes provided these procedures have been conducted as specified in the protocol.
2. Age ≥ 18 years.
3. Diagnosis of pancreatic islet cell tumors, well differentiated gastrointestinal NETs, pulmonary carcinoids and well differentiated thymic carcinoids. Locally-advanced or metastatic disease documented as progressive by CT scan, MRI, or Octreoscan at baseline and within 12 months prior to baseline. The previous scans will be used to classify the patient as having progressive disease at baseline according to RECIST criteria. Octreoscan results may be used to document progressive disease at baseline, but not for RECIST determination during the study.
4. ECOG performance status 0-1.
5. Disease not amenable to surgery, radiation or combined modality therapy with curative intent.
6. Presence of at least one dimensionally measurable target lesion for further evaluation according to RECIST 1.0 criteria (contrast enhancing lesion with the largest diameter > 1cm, based on CT or MRI scan done within 4 weeks before the start of treatment).
7. Patients could have received treatment with somatostatin analogs, chemotherapy, anti-VEGF, and anti-mTOR agents previously to the entrance into this study if the final toxicity was grade ≤ 1.
8. From patients who sign an informed consent form to donate biological samples: Tumor tissue must be provided for all available subjects at baseline and serum samples will be collected at baseline and at week 12 of treatment for biomarker analysis as defined at the biomarker section of this protocol.
9. Adequate organ system function as follows:

   9.1.Hematologic system:
   * Absolute neutrophil count (ANC) ≥ 1.5 X 10^9/L
   * Hemoglobin (1) ≥ 9 g/dL (5.6 mmol/L)
   * Platelets ≥ 100 X 10^9/L
   * Prothrombin time (PT) or international normalized ratio (INR) ≤ 1.2 X upper limit of normal (ULN)
   * Partial thromboplastin time (PTT) ≤ 1.2 X ULN

   9.2.Hepatic system (2):
   * Total bilirubin ≤ 1.5 X ULN
   * AST and ALT ≤ 2.5 X ULN

   9.3.Renal system:
   * Serum creatinine ≤ 1.5 mg/dL (133 µmol/L),

   Or, if greater than 1.5 mg/dL:
   * Calculated creatinine clearance ≥ 50 mL/min

   (Note 1):"Subjects should not have had a transfusion within 7 days of screening assessment." (Note 2): "Concomitant elevations in bilirubin and AST/ALT above 1.0 x ULN are not permitted"
10. A female is eligible to enter and participate in this study if she is of:

    10.1.Non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who has had:
    * A hysterectomy
    * A bilateral oophorectomy (ovariectomy)
    * A bilateral tubal ligation
    * Is post-menopausal

    10.2.Childbearing potential, including any female who has had a negative serum pregnancy test within 2 weeks prior to the first dose of study treatment, preferably as close to the first dose as possible, and agrees to use adequate contraception. GETNE acceptable contraceptive methods, when used consistently and in accordance with both the product label and the instructions of the physician, are as follow:
    * An intrauterine device with a documented failure rate of less than 1% per year.
    * Vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
    * Complete abstinence from sexual intercourse for 14 days before exposure to investigational product, through the dosing period, and for at least 21 days after the last dose of investigational product.
    * Double-barrier contraception (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide).
    * Oral contraceptives
    * Female subjects who are lactating should discontinue nursing prior to the first dose of study drug and should refrain from nursing throughout the treatment period and for 14 days following the last dose of study drug.
11. Life expectancy > 3 months.
12. Able to swallow oral compound.
13. Signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial prior to enrollment.
14. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.

Exclusion Criteria:

1. Diagnosis of any second malignancy within the last 5 years, except for adequately treated basal cell or squamous cell skin cancer, or in situ carcinoma of the cervix uteri.
2. History or clinical evidence of central nervous system (CNS) metastases or leptomeningeal carcinomatosis, except for individuals who have previously-treated CNS metastases, are asymptomatic, and have had no requirement for steroids or anti-seizure medication for 6 months prior to first dose of study drug. Screening with CNS imaging studies (computed tomography [CT] or magnetic resonance imaging [MRI]) is required only if clinically indicated or if the subject has a history of CNS metastases.
3. Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

   3.1.Active peptic ulcer disease 3.2.Known intraluminal metastatic lesion/s with risk of bleeding 3.3.Inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease), or other gastrointestinal conditions with increased risk of perforation 3.4.History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
4. Clinically significant gastrointestinal abnormalities that may affect absorption of investigational product including, but not limited to:

   4.1.Malabsorption syndrome 4.2.Major resection of the stomach or small bowel. 4.3.Active peptic ulcer disease 4.4.Known intraluminal metastatic lesion/s with risk of bleeding 4.5.Inflammatory bowel disease (e.g. ulcerative colitis, Chrohn's disease), or other gastrointestinal conditions with increased risk of perforation 4.6.History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days prior to beginning study treatment.
5. Presence of uncontrolled infection.
6. Corrected QT interval (QTc) > 480 msecs using Bazett's formula.
7. History of any one or more of the following cardiovascular conditions within the past 6 months:

   7.1.Cardiac angioplasty or stenting 7.2.Myocardial infarction 7.3.Unstable angina 7.4.Coronary artery bypass graft surgery 7.5.Symptomatic peripheral vascular disease 7.6.Class III or IV congestive heart failure, as defined by the New York Heart Association (NYHA)
8. Poorly controlled hypertension [defined as systolic blood pressure (SBP) of ≥140 mmHg or diastolic blood pressure (DBP) of ≥ 90mmHg].
9. History of cerebrovascular accident including transient ischemic attack (TIA), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months.

   Note: Subjects with recent DVT who have been treated with therapeutic anti-coagulating agents for at least 6 weeks are eligible.
10. Prior major surgery or trauma within 28 days prior to first dose of study drug and/or presence of any non-healing wound, fracture, or ulcer (procedures such as catheter placement not considered to be major).
11. Evidence of active bleeding or bleeding diathesis.
12. Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels.
13. Hemoptysis in excess of 2.5ml within 8 weeks of first dose of study drug.
14. Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures.
15. Unable or unwilling to discontinue use of prohibited medications list in Concomitant Medication Section for at least 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.
16. Treatment with any of the following anti-cancer therapies:

    * radiation therapy, surgery or tumor embolization within 28 days prior to the first dose of pazopanib, or
    * chemotherapy, immunotherapy, biological therapy, investigational therapy or hormonal therapy within 28 days prior to the first dose of pazopanib.
17. Any ongoing toxicity from prior anti-cancer therapy that is > Grade 1 and/or that is progressing in severity, except alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-01-26 (Actual); Primary Completion 2013-04 (Actual); Study Completion 2015-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Grande Pulido, MD, Study Chair — Grupo Espanol de Tumores Neuroendocrinos
Locations (10):
- Spain (10):
  - Institut Català d'Oncologia L'Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Centro Integral Oncológico Clara Campal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitari Son Espases, Palma de Mallorca
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza

REFERENCES:
- [Derived] Grande E, Capdevila J, Castellano D, Teule A, Duran I, Fuster J, Sevilla I, Escudero P, Sastre J, Garcia-Donas J, Casanovas O, Earl J, Ortega L, Apellaniz-Ruiz M, Rodriguez-Antona C, Alonso-Gordoa T, Diez JJ, Carrato A, Garcia-Carbonero R. Pazopanib in pretreated advanced neuroendocrine tumors: a phase II, open-label trial of the Spanish Task Force Group for Neuroendocrine Tumors (GETNE). Ann Oncol. 2015 Sep;26(9):1987-1993. doi: 10.1093/annonc/mdv252. Epub 2015 Jun 10. PMID 26063633

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between January 2011 and March 2012, a total of 44 patients were enrolled at 9 Spanish sites, belonging to Group for Neuroendocrine Tumors (GETNE).
Groups:
- Arm of Pazopanib: Single arm of pazopanib 800 mg, administered once a day as the only treatment.
Period: Overall Study
Arm/Group | Arm of Pazopanib
Started | 44
Completed | 44
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Arm of Pazopanib
Number analyzed (Participants) | 44
Age, Continuous [Mean (Full Range); unit: years] | 60 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 44
Tumor type [Count of Participants; unit: Participants]
  Pancreatic islet cell tumors | 18
  Gastrointestinal neuroendocrine tumors | 15
  Pulmonary carcinoid tumors | 5
  Thymic carcinoid tumors | 3
  Unknown primary origin tumors | 3
Functional tumor status [Number; unit: participants] — Nonfunctional tumors-no specific clinical syndrome is observed; Functional tumors-the tumors' secretions lead to clinical symptoms.
  participants
    Functional | 13
    Nonfunctional | 31
Histologic status of tumor [Count of Participants; unit: Participants]
  Well differentiated | 30
  Moderately differentiated | 3
  Poorly differentiated | 2
  Unknown | 9
Ki67 index [Number; unit: participants]
  ≤2% | 6
  3%-10% | 13
  >10% | 5
  Unknown | 20
Previous biologic treatment [Count of Participants; unit: Participants]
  Everolimus | 11
  Multitargeted agent | 16
  mTOR and multitargeted inhibitor | 8
  None | 9
Previous chemotherapy [Count of Participants; unit: Participants] | 16
Previous somatostatin analogs [Count of Participants; unit: Participants] | 35
Concurrent somatostatin analogs [Count of Participants; unit: Participants] | 30

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate
Description: Per Response Evaluation Criteria In Solid Tumor Criteria (RECIST v1.0) for target lesions and assessed by MRI: complete response (CR) considered as dissapereance of all target lesions: partial response (PR), considered as >=30% decrease in the sum of the longest diameter of target lesions, or stable disease (SD) considered as a decrease <30%, after pazopanib was started. Clinical benefit rate (CBR) was defined as the percentage of patients achieving CR, PR or SD.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm of Pazopanib
Number analyzed (Participants) | 15
Participants | 11

2. Secondary Outcome: Number of Patients Who Had an Event (Disease Progression or Death)
Description: Per Response Evaluation Criteria In Solid Tumor Criteria (RECIST v1.0) for target lesions and assessed by MRI, considered as the proportion of patietnts whose target lesions have been reported with a >=30% increase in the sum of the longest diameter of target lesions.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm of Pazopanib
Number analyzed (Participants) | 40
Participants | 35

3. Secondary Outcome: Radiological Objective Complete Response Rate
Description: Per Response Evaluation Criteria In Solid Tumor Criteria (RECIST v1.0) for target lesions and assessed by MRI, considered as the proportion of patients whose target lessions have dissaperead after treatment.
Time Frame: 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm of Pazopanib
Number analyzed (Participants) | 44
Participants | 4

4. Secondary Outcome: Duration of Response (DoR)
Description: Defined, for the subset of patients with a confirmed CR o PR, as the time from first documented evidence of CR or PR until first documented disease progression or death due to any cause. The DR data will be censored the day after the last evaluation in those patients who did not present an objective tumoral progression and did not died during their participation in the trial. The DR will be assessed only in the subset of patients presenting objective response.
Time Frame: 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm of Pazopanib
Number analyzed (Participants) | 44
months | 11.3 [2.0 to 20.6]

5. Secondary Outcome: Safety Assessment Criteria
Description: Security and tolerance to the study medication will be determined evaluating the type, incidence, severity, timing, seriousness and connections with the treatment of the reported adverse events, physical examinations and laboratory tests. Toxicity will be classified according to NCI-CTCAE v 4.0.
Time Frame: 3 years
Population: Number of participantes with grade 3 or 4 AEs
Measure: Count of Participants; unit: Participants
Arm/Group | Arm of Pazopanib
Number analyzed (Participants) | 44
Participants | 28

6. Secondary Outcome: Predictive Value of Baseline CTC (Count of 0) for Response to Treatma
Description: Predictive value of the differente biomarkers included in the study was evaluated using multivariate analysis.
Time Frame: 3 years
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | Arm of Pazopanib
Number analyzed (Participants) | 44
Odds ratio | 6.2 [0.45 to 86.5]

ADVERSE EVENTS:
Time Frame: 4 years, 8 months
Arm/Group | Arm of Pazopanib
All-Cause Mortality (participants affected / at risk) | 1/44
Serious Adverse Events (participants affected / at risk) | 19/44
Other Adverse Events (participants affected / at risk) | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm of Pazopanib (N=44)
HEPATOTOXICITY (Hepatobiliary disorders) | 1 (1)
DIABETIC DECOMPENSATION (Endocrine disorders) | 1 (1)
INTESTINAL SUBOCLUSION (Gastrointestinal disorders) | 1 (1)
HYPERGLUCEMIA (Metabolism and nutrition disorders) | 1 (1)
GENERALIZED CRISIS (Psychiatric disorders) | 1 (1)
OBSTRUCTIVE ICTERY (Hepatobiliary disorders) | 1 (1)
OLIGOARTRALGIAS (Musculoskeletal and connective tissue disorders) | 1 (1)
HYPERTENSIVE CRISIS (Vascular disorders) | 1 (1)
RESPIRATORY INFECTION BY E.COLI (Infections and infestations) | 1 (1)
ACTIVE TUBERCULOSIS (Infections and infestations) | 1 (1)
CEREBELLY HEMATOMY (Vascular disorders) | 1 (1)
ALT AND AST INCREASE (Hepatobiliary disorders) | 1 (1)
CELLULITIS (Skin and subcutaneous tissue disorders) | 1 (1)
DISSEMINATED INTRAVASCULAR COAGULATION (Vascular disorders) | 1 (1)
COLANGITIS (Hepatobiliary disorders) | 1 (3)
COMA HYPOGLYCEMIC (Metabolism and nutrition disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
ABDOMINAL PAIN (General disorders) | 1 (1)
TUMORAL PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
HEPATIC ENCEPHALOPATHY (Hepatobiliary disorders) | 1 (1)
BILIARY STENOSIS (Hepatobiliary disorders) | 1 (1)
HYPERTRANSAMINASEMIA (Hepatobiliary disorders) | 1 (1)
LIVER FAILURE (Hepatobiliary disorders) | 1 (1)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 1 (1)
INJURY IN HYPOPHYSIS (Injury, poisoning and procedural complications) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 2 (4)
PROGRESSION DISEASE (General disorders) | 1 (1)
INTESTINAL BLEEDING (Gastrointestinal disorders) | 1 (1)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Small sample size, heterogeneous location and degree of differentiation of primary tumors, and lack of an appropriate control group. Additionally,response was evaluated by the investigator and not by an independent committee.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No